CLINICAL TRIAL: NCT03146169
Title: Training Program for Community Health Campaign: Fitter Families Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Research Officer, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UW15 - 401
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Motor Activity
MeSH Terms: conditions — Motor Activity | interventions — Sensitivity Training Groups

STUDY DESIGN:
Intervention Model Description: A four-session training workshop is provided to the trainees in order to enhance their competence and performance for conducing and/or assisting the implementation of community -based interventions and activities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training group (Experimental): Four two-hour training sessions were conducted at baseline, and one week, one month and three months after the first session.
  Interventions: Behavioral: Training group

INTERVENTIONS:
Behavioral: Training group — The training workshop includes four two-hour sessions:
  Session one - a knowledge, self-efficacy, and motivation enhancement session at baseline; Session two - an interpersonal communication and leadership skills session at one week; Session three - a motivation enhancement session at one month Session four - an experience sharing session at three months

SUMMARY:
In recent years, Hong Kong has been undergoing rapid changes with macro social and economic trends. The increasingly complex and diverse family structure contribute to concerns regarding the well-being of families in Hong Kong, including their health, happiness and harmony (FAMILY 3Hs). Family life and health education should be strengthened to meet the increasing needs of promoting healthy active lifestyle among Hong Kong families. In this connection, the FAMILY Project initiates the Fitter Families Project (FFP) with a focus on "FAMILY Holistic Health", will be conducted in order to increase the awareness of the importance of FAMILY 3Hs. FFP is a community-based research project with 3 main components - train-the-trainer program, community-based family interventions and public education events. It is expected that trainees from the train-the-trainer program will acquire adequate skills to organize community-based health education programs effectively. Participants of the community-based family interventions will gain knowledge on family holistic health and live a healthy active lifestyle. Attendees of the public education events will become more aware of the importance of FAMILY 3Hs.

DETAILED DESCRIPTION:
In 2011, United Nations (UN) addressed the prevention and control of four non-communicable diseases (NCDs: cancer, cardiovascular disease, chronic respiratory disease, and diabetes mellitus) worldwide. The UN, in its Political Declaration, recognized the critical importance of reducing the exposure to the common modifiable risk factors for NCDs, namely, tobacco use, unhealthy diet, physical inactivity, and the harmful use of alcohol.In Hong Kong, NCDs are responsible for more than 85% of all deaths and most of these are preventable. FAMILY Project Cohort Study (2014) also found that 88.6% of Hong Kong people had inadequate vegetable and fruit intake, 70.6% had inadequate physical exercise, 26.4% were overweight and 5.4% were obese.

Families worldwide have been undergoing rapid changes with macro, social and economic trends. Demographic shifts, economic upheavals, changing societal norms and values, immigration across national borders and migration within nations are creating new and altered structures, processes and relationships within families. The increasingly complex and diverse family structure contributes to concerns regarding the well-being of families in Hong Kong, including their health, happiness and harmony (FAMILY 3Hs). Family life and health education should be strengthened to meet the increasing needs of promoting healthy lifestyle among Hong Kong families.

The Fitter Families Project is developed based on the strong foundation of the Learning Families Project in the previous years. In view of the health challenges locally and globally, the new phase of FAMILY project will put more emphasis on health in the upcoming three years. Following the themes on FAMILY health, happiness and harmony (3Hs), the Fitter Families Project focuses on family holistic health with emphasis on the interaction and integration of both physical and psychosocial health.

As an initial step of this project, the investigators conducted a need assessments before designing and conducting a train-the-trainer program. The train-the-trainer program aimed to prepare the staff and lay volunteers to conduct and or assist to implement a series of community-based activities and interventions for the participants of Fitter Families Project. Focus group interviews were conducted to obtain feedback and opinion from the trainees . Questionnaire assessments were conducted before, immediately after finishing the training, three months after training.

ELIGIBILITY:
Inclusion Criteria:

* Chinese speaking
* able to complete assessments

Exclusion Criteria:

* not fit the inclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in trainees' learning | baseline, immediately after first session "up to 30 min", one month and three months
  Assessed by outcome-based questionnaire

SECONDARY OUTCOMES:
Trainees' reactions to training content | Immediately after the training workshop
  Assessed by outcome-based questionnaire
Trainees' changes in the frequency and amount on performing physical exercise adn Zero Time Exercise | baseline, one month and three months
  Assessed by outcome-based questionnaire on performing moderate exercise, vigorous exercise and Zero Time Exercise and walking
Trainees' changes in grip strength (kg) | baseline and one month
  assessed by a hand grip dynamometer
Trainees' changes in chair stand (times) | Assessed 30s Chair stand test ( a test counting number of times from sitting position to standing position in 30 seconds
  baseline and one month
Trainees' changes in single-leg standing time (second) | Assessed by a single-leg stance test ( a test measuring the longest duration of a single leg in 120 seconds)
  baseline and one month
Trainees' changes in seat and reach (cm) | Baseline and one month
  Assessed by a ruler
Trainees' changes in body fat (%) | Baseline and one month
  Assessed by a standard body fat and weight measuring scale
Trainees' changes in body weight (kg) | Baseline and one month
  Assessed by a standard body fat and weight measuring scale
Trainees' changes in frequency and amount on performing physical activity and Zero Time Exercise) | baseline, one month and three months
  Assessed by outcome-based questionnaire on performing moderate exercise, vigorous exercise and Zero Time Exercise and walking
Trainees' changes in personal happiness | baseline, one month and three months
  Assessed by outcome-based questionnaire
Trainees' changes in personal health | baseline, one month and three months
  Assessed by outcome-based questionnaire
Trainees' changes in family health | baseline, one month and three months
  Assessed by outcome-based questionnaire
Trainees' changes in family happiness | baseline, one month and three months
  Assessed by outcome-based questionnaire
Trainees' changes in family harmony | baseline, one month and three months
  Assessed by outcome-based questionnaire
Trainees' changes in sharing health knowledge with family members in relation to physical activity | baseline, one month and three months
  Assessed by outcome-based questionnaire
Trainees' changes in doing physical activity and exercise with family | baseline, one month and three months
  Assessed by outcome-based questionnaire
Trainees' comments on the received electronic health messages | baseline, one month and three months
  Assessed by outcome-based questionnaire
Community participants' changes in family health | baseline, one month and three months
  Assessed by outcome-based questionnaire
Community participants' changes in family happiness | baseline, one month and three months
  Assessed by outcome-based questionnaire
Community participants' changes in family harmony | baseline, one month and three months
  Assessed by outcome-based questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Agnes YK Lai, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Christian Family Service Centre, Kwun Tong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The minimal anonymized dataset will be available upon request to interested researchers. For interested researchers, please contact, Ms Grace Lau (email gclau@hku.hk), (School of Public Health, The University of Hong Kong) for further information."

REFERENCES:
- [Background] Wacharasin C, Theinpichet S. Family nursing practice, education, and research: what is happening in Thailand? J Fam Nurs. 2008 Nov;14(4):429-35. doi: 10.1177/1074840708327515. PMID 19139157
- [Background] Denham SA. Family routines: a structural perspective for viewing family health. ANS Adv Nurs Sci. 2002 Jun;24(4):60-74. doi: 10.1097/00012272-200206000-00010. PMID 12699277
- [Background] Yoshikawa H. Integrating methods in the science of family health: new directions from an institute of medicine workshop report. Arch Pediatr Adolesc Med. 2012 Jul 1;166(7):659-61. doi: 10.1001/archpediatrics.2012.510. No abstract available. PMID 22751883
- [Background] Anderson KH, Tomlinson PS. The family health system as an emerging paradigmatic view for nursing. Image J Nurs Sch. 1992 Spring;24(1):57-63. doi: 10.1111/j.1547-5069.1992.tb00700.x. PMID 1541473
- [Derived] Lai AYK, Stewart SM, Wan ANT, Shen C, Ng CKK, Kwok LT, Chan SS, Ho DSY, Lam TH. Training to implement a community program has positive effects on health promoters: JC FAMILY Project. Transl Behav Med. 2018 Nov 21;8(6):838-850. doi: 10.1093/tbm/iby070. PMID 29961808